CLINICAL TRIAL: NCT07086079
Title: A Clinical Study to Evaluate the Breast Milk and Plasma Pharmacokinetics of MK-8591A in Healthy Lactating Female Participants
Brief Title: A Study of Doravirine/Islatravir in Healthy Lactating Females (MK-8591A-061)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8591A-061; MK-8591A-061 (Other: MSD)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DOR/ISL (Experimental): Participants will receive DOR/ISL as an oral fixed-dose combination tablet once daily on Days 1 to 7.
  Interventions: Drug: DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — Oral tablet
  Other Names: MK-8591A

SUMMARY:
The goal of this study is to learn what happens to doravirine (DOR) and islatravir (ISL) in a healthy lactating female's body over time. Researchers want to learn if DOR and ISL are in breast milk.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is at least 6-weeks postpartum at the time of administration of study drug, following the delivery of a healthy singleton neonate
* Is willing and able to express breast milk using an electric pump prior to study drug administration and is expected to be able to express at least 4 times over a 24-hour period after study drug administration

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, psychiatric, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has had mastitis within 30 days prior to administration of study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy Lactating Female Participants
Enrollment: 12 (Actual)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative Amount of DOR Excreted in Breast Milk From 0 to 24 Hours (Ae0-24hrs) | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the Ae0-24hrs after administration of DOR.
Body Weight Normalized Infant Theoretical Dose of DOR | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to calculate the theoretical daily (24 hour) infant dose of DOR as normalized by participant-reported infant body weight.
Relative Infant Theoretical Dose of DOR | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to calculate the theoretical daily (24 hour) infant dose of DOR relative to the maternal dose.
Cumulative Amount of Total ISL Excreted in Breast Milk From 0 to 24 Hours (Ae0-24hrs) | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the Ae0-24hrs after administration of total ISL.
Body Weight Normalized Infant Theoretical Dose of ISL | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to calculate the theoretical daily (24 hour) infant dose of ISL as normalized by participant-reported infant body weight.
Relative Infant Theoretical Dose of ISL | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to calculate the theoretical daily (24 hour) infant dose of ISL relative to the maternal dose.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From 0 to 24 Hours (AUC0-24hrs) of DOR in Breast Milk | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the AUC0-24hrs of DOR.
Maximum Concentration (Cmax) of DOR in Breast Milk | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the Cmax of DOR.
Time to Maximum Concentration (Tmax) of DOR in Breast Milk | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the Tmax of DOR
AUC0-24hrs of Total ISL in Breast Milk | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the AUC0-24hrs of total ISL.
Cmax of Total ISL in Breast Milk | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the Cmax of total ISL.
Tmax of Total ISL in Breast Milk | Predose and at designated timepoints up to 24 hours postdose
  Breast milk samples will be collected to determine the Tmax of total ISL.
AUC0-24hrs of DOR in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the AUC0-24hrs of DOR.
Cmax of DOR in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the Cmax of DOR.
Tmax of DOR in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the Tmax of DOR.
Concentration at 24 Hours (C24) of DOR in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the C24 of DOR.
AUC0-24hrs of ISL in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the AUC0-24hrs of ISL.
Cmax of ISL in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the Cmax of ISL.
Tmax of ISL in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the Tmax of ISL.
C24 of ISL in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Plasma samples will be collected to determine the C24 of ISL.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS Missouri ( Site 0001), Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com